CLINICAL TRIAL: NCT00362427
Title: A Randomized Trial to Assess the Immunogenicity and Safety of PR5I With an Adjuvant Composition Enhancement to the Hepatitis B Component and When Given Concomitantly With Prevnar®
Brief Title: Study of PR5I, a Pediatric Combination Vaccine With Enhanced Hepatitis B Component Given Concomitantly With Prevnar®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR504
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Diphtheria; Pertussis; Polio; Hepatitis B; Tetanus
Keywords: Hepatitis B; Pertussis; Diphtheria; Tetanus; H. influenzae type b; Polio
MeSH Terms: conditions — Diphtheria; Whooping Cough; Poliomyelitis; Hepatitis B; Tetanus; Haemophilus Infections | interventions — Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine; pentacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: Hybrid 5 component DTaP, Vero IPV, Hep B and PRP-OMPC
- Group B (Experimental)
  Interventions: Biological: Hybrid 5 component DTaP, Vero IPV, Hep B and PRP-OMPC
- Group C (Active Comparator)
  Interventions: Biological: Hybrid 5 component DTaP, Vero IPV, Hep B and PRP-OMPC

INTERVENTIONS:
Biological: Hybrid 5 component DTaP, Vero IPV, Hep B and PRP-OMPC — 0.5 mL, 4 doses, IM
  Other Names: PR5I
  Arms: Group A
Biological: Hybrid 5 component DTaP, Vero IPV, Hep B and PRP-OMPC — 0.5 Ml, 4 doses, IM
  Other Names: PR5I
  Arms: Group B
Biological: Hybrid 5 component DTaP, Vero IPV, Hep B and PRP-OMPC — 0.5 mL, 4 doses, IM with concommitant vaccines
  Other Names: PR5I; PENTACEL™; NGERIX-B®
  Arms: Group C

SUMMARY:
PR5I, a hexavalent pediatric combination vaccine is being developed to reduce the number of injections during the first 2 years of life while providing a complete course of immunization against infection caused by H. influenzae type b, hepatitis B virus, Corynebacterium diphtheriae, Clostridium tetani, Bordetella pertussis, and poliovirus types 1, 2, and 3.

Primary Objective: To evaluate immunogenicity of PR5I with the adjuvant composition enhancement to the hepatitis B component when administered concomitantly with Prevnar®

Secondary Objectives: To assess the safety and immunogenicity of PR5I when administered concomitantly, or one month apart with Prevnar® or separately with licensed vaccines used for routine infant vaccination in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 42 to 89 days inclusive on the day of inclusion.
* Born at full term of pregnancy (>37 weeks).
* Informed consent form signed by the parent(s) or legally authorized representative.
* Able to attend all scheduled visits and to comply with the study procedures.
* Parent or legally authorized representative has access to a telephone.
* Parent or legally authorized representative able to read and write in English or French.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Personal or immediate family history of congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy.
* Known or suspected systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances as the trial vaccine(s).
* Chronic illness that could interfere with trial conduct or completion.
* Received blood or blood-derived products since birth.
* Any vaccination preceding the first trial vaccination or planned in the 4 weeks after any trial vaccination (flu vaccine may be given a minimum of 4 weeks prior to the first study vaccination).
* Previous vaccination with any acellular pertussis- (DTaP) or whole cell pertussis- (DTwP) based combination vaccines, Haemophilus influenzae type b (Hib)-conjugate, poliovirus, hepatitis B, or pneumococcal conjugate vaccines.
* Coagulation disorder contraindicating IM vaccination.
* Clinically significant findings on review of systems (determined by investigator or sub-investigator to be sufficient for exclusion).
* Developmental delay or neurological disorder.
* Any condition which, in the opinion of the investigator, would interfere with the evaluation of the vaccine or pose a health risk to the subject.
* Documented Hepatitis B surface Antigen (HBsAg) seropositivity in the child or his/her mother.
* History of Hib, hepatitis B, diphtheria, tetanus, pertussis or poliovirus disease.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 460 (Actual)
Dates: Start 2006-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immune response of subjects that received PR5I concomitantly with Prevnar | 14 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (7):
- Canada (7):
  - Coquitlam, British Columbia
  - Surrey, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Ottawa, Ontario
  - Beauport, Quebec
  - Montreal, Quebec

REFERENCES:
- [Derived] Halperin SA, Tapiero B, Dionne M, Meekison W, Diaz-Mitoma F, Zickler P, Rubin E, Embree J, Bhuyan P, Lee A, Li M, Tomovici A. Safety and immunogenicity of a toddler dose following an infant series of a hexavalent diphtheria, tetanus, acellular pertussis, inactivated poliovirus, Haemophilus influenzae type b, hepatitis B vaccine administered concurrently or at separate visits with a heptavalent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2014 Jan;33(1):73-80. doi: 10.1097/01.inf.0000437806.76221.20. PMID 24346596
- [Derived] Tapiero B, Halperin SA, Dionne M, Meekison W, Diaz-Mitoma F, Zickler P, Rubin E, Embree J, Bhuyan P, Lee AW, Li M, Tomovici A. Safety and immunogenicity of a hexavalent vaccine administered at 2, 4 and 6 months of age with or without a heptavalent pneumococcal conjugate vaccine: a randomized, open-label study. Pediatr Infect Dis J. 2013 Jan;32(1):54-61. doi: 10.1097/INF.0b013e3182717edf. PMID 23241989
- See also: Related Info — http://www.sanofipasteur.com